CLINICAL TRIAL: NCT01636245
Title: Immunogenicity and Safety of Three Consecutive Lots of a New Inactivated Enterovirus Type 71 (EV71) Vaccine: A Double-blind, Randomized and Controlled Trial
Brief Title: Immunogenicity and Safety of Three Consecutive Lots of a New Inactivated Enterovirus Type 71 (EV71) Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PRO-EV71-3002
Record Dates: First submitted 2012-07-05; First posted 2012-07-10 (Estimated); Last update posted 2013-03-15 (Estimated); Status verified 2013-03

CONDITIONS: Hand, Foot and Mouth Disease
Keywords: 71 vaccine; HFMD; consistency of three consecutive lots; immunogenicity
MeSH Terms: conditions — Hand, Foot and Mouth Disease | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Lot 1 (Experimental): inactivated vaccine (Lot 1) against EV71 of 400U /0.5ml in 350 infants aged 6 months to 5 years old on day 0,28
  Interventions: Biological: three consecutive lots of EV71 vaccine
- Lot 2 (Experimental): inactivated vaccine (Lot 2) against EV71 of 400U /0.5ml in 350 infants aged 6 months to 5 years old on day 0,28
  Interventions: Biological: three consecutive lots of EV71 vaccine
- Lot 3 (Experimental): inactivated vaccine (Lot 3) against EV71 of 400U /0.5ml in 350 infants aged 6 months to 5 years old on day 0,28
  Interventions: Biological: three consecutive lots of EV71 vaccine
- Placebo (Placebo Comparator): Placebo in 350 infants aged 6 months to 5 years old on day 0,28
  Interventions: Biological: placebo

INTERVENTIONS:
Biological: three consecutive lots of EV71 vaccine — inactivated vaccine (vero cell) against EV71 of 400U /0.5ml, two doses, 28 days interval
  Other Names: Vaccine groups
  Arms: Lot 1; Lot 2; Lot 3
Biological: placebo — placebo, two doses, 28 days interval
  Other Names: Control group
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the immunogenicity and safety of three consecutive lots of EV71 Vaccines in healthy infants volunteers aged from 6 months to 5 years old.

DETAILED DESCRIPTION:
The data from the phase I and II study suggested that the inactivated EV71 vaccine (vero cell) had a clinically acceptable safety and good immunogenicity for healthy Chinese infants. The phase III study of inactivated vaccine has initiated on Jan 2012 in China. Over 10,000 healthy infants have revieved the vaccines and no unexpected severe adverse reactions were reported. According to the requirement of SFDA (China), the sponsor should also provide the evidence for the consistency of three consecutive lots of EV71 Vaccines before the application for the market. Thus, a clinical trial to evaluate the immunogenicity and safety of three consecutive lots of EV71 Vaccines in healthy infants volunteers is planed to conduct.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females, aged from 6 months to 11 years old Health is determined by medical history, physical examination, laboratory examination and clinical judgment of the investigator
* Provided legal identification for the sake of recruitment
* Subjects and/or parent(s)/legal guardian(s) are able to understand and sign informed consents

Exclusion Criteria:

* History of Hand-foot-mouth Disease
* Subject that has allergic history of vaccine, or allergic to any ingredient of vaccine
* Serious adverse reactions to vaccines such as anaphylaxis, hives, respiratory difficulty, angioedema, or abdominal pain
* Congenital malformations or developmental disorders, genetic defects, or severe malnutrition
* Epilepsy, seizures or convulsions history, or family history of mental illness
* Autoimmune disease or immunodeficiency, or parents, brothers and sisters have autoimmune diseases or immunodeficiency
* History of asthma, angioedema, diabetes or malignancy
* History of thyroidectomy or thyroid disease that required medication within the past 12 months
* Bleeding disorder diagnosed by a doctor (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws
* Asplenia, functional asplenia or any condition resulting in the absence or removal the spleen
* Acute illness or acute exacerbation of chronic disease within the past 7 days
* Any history of immunosuppressive medications or cytotoxic medications or inhaled corticosteroids within the past six months (with the exception of corticosteroid nasal spray for allergic rhinitis or topical corticosteroids for an acute uncomplicated dermatitis)
* History of any blood products within 3 months
* Administration of any live attenuated vaccine within 14 days
* Administration of subunit or inactivated vaccines ,e.g., pneumococcal vaccine, or allergy treatment within 7 days
* Axillary temperature > 37.0 centigrade before vaccination
* Abnormal laboratory parameters before vaccination
* Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a volunteer's ability to give informed consent

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1400 (Actual)
Dates: Start 2012-07; Primary Completion 2012-09 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
The GMT of anti-EV71 antibodies in serum 28 days after the two-dose regimen | 28 days after first vaccination
  to evaluate the immunogenicity of anti-EV71 antibodies in serum 28 days after second vaccination

SECONDARY OUTCOMES:
Frequency of systemic and local adverse reactions after the first vaccination | 28 days after the first vaccination
  Frequency of systemic and local adverse reactions in healthy infants following first doses of EV71 vaccine
Frequency of systemic and local adverse reactions after the second vaccination | 28 days after the second vaccination
  Frequency of systemic and local adverse reactions in healthy infants following second doses of EV71 vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Yue-Mei Hu, BS, Principal Investigator — Jiangsu Center for Diseases Control and Prevention
Locations (1):
- Jurong, Zhenjiang, Jiangsu, China

REFERENCES:
- [Derived] Zhang H, An D, Liu W, Mao Q, Jin J, Xu L, Sun S, Jiang L, Li X, Shao J, Ma H, Huang X, Guo S, Chen H, Cheng T, Yang L, Su W, Kong W, Liang Z, Jiang C. Analysis of cross-reactive neutralizing antibodies in human HFMD serum with an EV71 pseudovirus-based assay. PLoS One. 2014 Jun 25;9(6):e100545. doi: 10.1371/journal.pone.0100545. eCollection 2014. PMID 24964084
- [Derived] Hu YM, Wang X, Wang JZ, Wang L, Zhang YJ, Chang L, Liang ZL, Xia JL, Dai QG, Hu YL, Mao QY, Zhu FC, Song YF, Gao F, Chen JT. Immunogenicity, safety, and lot consistency of a novel inactivated enterovirus 71 vaccine in Chinese children aged 6 to 59 months. Clin Vaccine Immunol. 2013 Dec;20(12):1805-11. doi: 10.1128/CVI.00491-13. Epub 2013 Oct 9. PMID 24108780